CLINICAL TRIAL: NCT07388901
Title: Randomized Controlled Trial of iRoot SP (Injectable Root Canal Sealer Paste) and nRoot SP (ENPUNUO Root Canal Sealer Paste) in Patients With Chronic Apical Periodontitis
Brief Title: In Vivo Study on the Material Properties of iRoot SP and nRoot SP Root Canal Sealers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Dental Hospital of Zhejiang University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2025-064
Record Dates: First submitted 2026-01-20; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Chronic Apical Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iRoot SP (Active Comparator): iRoot SP was used as the root canal sealer material during the root canal filling step of the root canal treatment.
  Interventions: Device: iRoot SP
- nRoot SP (Experimental): nRoot SP was used as the root canal sealer material during the root canal filling step of the root canal treatment.
  Interventions: Device: nRoot SP

INTERVENTIONS:
Device: iRoot SP — use iRoot SP in root canal treatment
  Arms: iRoot SP
Device: nRoot SP — use nRoot SP in root canal treatment
  Arms: nRoot SP

SUMMARY:
A randomized controlled trial was conducted to compare the treatment efficacy of iRoot SP and nRoot SP Root Canal Sealer Materials in patients with chronic apical periodontitis.

DETAILED DESCRIPTION:
This study aims to conduct a randomized controlled clinical trial to evaluate the 3-24months efficacy (including radiographic reduction of periapical radiolucency, postoperative pain, etc.) of the two materials in patients with chronic apical periodontitis. The objective is to provide evidence-based support for the optimization and clinical selection of domestically produced materials, thereby promoting the precise application of bioceramic sealers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Diagnosis of apical periodontitis conforming to the diagnostic criteria in Endodontics.
* The affected tooth is deemed restorable upon evaluation, with non-vital pulp requiring extirpation.
* The affected tooth is a single tooth with a fully developed apical foramen.
* No root resorption and no significant morphological variation of the root canal.
* The affected tooth is undergoing primary root canal treatment.
* Periapical radiolucency with a diameter of 1-5 mm and no peripheral sclerotic border observed on preoperative radiographs.
* Patient is in normal mental state, conscious, and capable of normal communication.
* Patient has provided informed consent.

Exclusion Criteria:

* Patients with alveolar bone loss exceeding one-third of the root length.
* Affected teeth with root fracture, root canal obstruction, calcification, or root surface caries.
* Patients with severe systemic diseases (e.g., osteoporosis, mental disorders, hepatic or renal insufficiency).
* Patients who have taken analgesics, immunosuppressants, or antibiotics within one week prior to enrollment.
* Patients with concurrent periapical cysts, oral tumors, or other oral diseases.
* Pregnant or lactating patients.
* Patients with dental phobia, severe gag reflex, limited mouth opening, or poor compliance.
* Patients with a known allergy to the root canal sealer materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
therapeutic effect | 3,6,12,24months
  Markedly Effective: Post-treatment X-ray examination shows complete resolution of the periapical radiolucency. The patient's chewing function is largely restored, and symptoms such as gingival swelling/pain, tooth discoloration, and occlusal discomfort have disappeared.
  Effective: Post-treatment X-ray examination shows significant reduction in the size of the radiolucency. The patient may experience mild percussion pain or discomfort. Chewing function is largely normal, and symptoms such as gingival swelling/pain, tooth discoloration, and occlusal discomfort show improvement.
  Ineffective: Post-treatment X-ray examination shows no reduction or even enlargement of the radiolucency. The patient reports significant percussion pain. Symptoms such as gingival swelling/pain, tooth discoloration, and occlusal discomfort show no improvement.

SECONDARY OUTCOMES:
clinical manifestation | 3,6,12,24months
  Four distinct clinical assessments to be evaluated at 3, 6, 12, and 24 months postoperatively: tooth mobility, assessed clinically using a standard grading scale (Miller index. Grade I: Mobility with a buccolingual displacement of ≤1 mm; Grade II: Mobility with a buccolingual displacement of 1-2 mm, possibly accompanied by slight mesiodistal mobility; Grade III: Mobility with a buccolingual or mesiodistal displacement exceeding 2 mm, or the presence of vertical mobility.) ; periodontal probing depth, measured at designated sites(mesiobuccal, midbuccal, distobuccal mesiolingual, midlingual, distolingual).) around the tooth with a periodontal probe and recorded in millimeters; percussion pain, evaluated by vertical and horizontal tapping and documented either as a binary presence/absence; the presence of a sinus tract, determined through visual inspection and verification with a gutta-percha point if necessary and recorded as a binary outcome. Each parameter will be analyzed independent
Imaging findings | 3,6,12,24months
  Change in the size of the periapical radiolucent area. Specifically, after acquiring the image, the DICOM format image will be imported into 3D slicer, the maximum diameter of the apical low-density shadow will be measured using the ruler function, the range of the apical low-density shadow will be divided using the segment editor module, and the volume of the periapical shadow will be calculated using the segment statistics module

CONTACTS AND LOCATIONS:
Overall Officials: Tu Yan, Principal Investigator — School of Stomatology, The Affiliated Stomatology Hospital of Zhejiang University School of Medicine
Locations (1):
- School of Stomatology, The Affiliated Stomatology Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang, China

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT07388901/Prot_SAP_000.pdf
  • Informed Consent Form (2025-05-31): https://cdn.clinicaltrials.gov/large-docs/01/NCT07388901/ICF_001.pdf